CLINICAL TRIAL: NCT06132958
Title: A Phase 3, Randomized, Active-controlled, Open-label, Multicenter Study to Compare the Efficacy and Safety of MK-2870 Monotherapy Versus Treatment of Physician's Choice in Participants With Endometrial Cancer Who Have Received Prior Platinum-based Chemotherapy and Immunotherapy (MK-2870-005/ENGOT-en23/GOG-3095)
Brief Title: Sacituzumab Tirumotecan (MK-2870) in Post Platinum and Post Immunotherapy Endometrial Cancer (MK-2870-005)
Acronym: TroFuse-005
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: European Network for Gynaecological Oncological Trial groups(ENGOT) (Unknown); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2870-005; 2023-504816-14-00 (Registry Identifier: EU CT); U1111-1288-7581 (Registry Identifier: UTN); jRCT2031240041 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Antibody-drug conjugate (ADC); Trophoblast cell-surface antigen 2 (TROP2)
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Doxorubicin; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab tirumotecan (Experimental): Participants will receive 4 mg/kg of sacituzumab tirumotecan via intravenous (IV) infusion on Day 1 of each 14-day cycle. Additionally, participants receive diphenhydramine (or equivalent), a Histamine (H2 antagonist) of investigator's choice, acetaminophen (or equivalent), and dexamethasone (or equivalent) per each drug's product label prior to the first 4 infusions of sacituzumab tirumotecan. At subsequent infusions, the H2 antagonist and dexamethasone are optional, at the discretion of the investigator.
  Interventions: Biological: Sacituzumab tirumotecan
- Chemotherapy (Active Comparator): Participants will receive 60 mg/m^2 of doxorubicin by IV infusion on Day 1 of each 21-day cycle; or 80 mg/m^2 of paclitaxel by IV infusion on Days 1, 8, and 15 of each 28-day cycle. Participants who experience either a severe hypersensitivity reaction to paclitaxel or an AE requiring discontinuation of paclitaxel may receive Nab-paclitaxel.
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — 4 mg/kg of sacituzumab tirumotecan by IV infusion
  Other Names: SKB264 MK-2870
  Arms: Sacituzumab tirumotecan
Drug: Doxorubicin — 60 mg/m^2 of doxorubicin by IV Infusion
  Other Names: ADRIAMYCIN®
  Arms: Chemotherapy
Drug: Paclitaxel — 80 mg/m^2 of paclitaxel by IV infusion
  Other Names: TAXOL®
  Arms: Chemotherapy
Drug: Nab-paclitaxel — 100 mg/m^2 of nab-paclitaxel by IV infusion
  Other Names: Abraxane
  Arms: Chemotherapy

SUMMARY:
Researchers are looking for new ways to treat people with endometrial cancer (EC) who have previously received treatment with platinum based therapy (a type of chemotherapy) and immunotherapy. Immunotherapy is a treatment that helps the immune system fight cancer. This clinical study will compare sacituzumab tirumotecan to chemotherapy. The goal of the study is to learn if people who receive sacituzumab tirumotecan live longer overall and without the cancer getting worse compared to people who receive chemotherapy.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has a histologically-confirmed diagnosis of endometrial carcinoma or carcinosarcoma.
* Has radiographically evaluable disease, either measurable or nonmeasurable per response evaluation criteria in solid tumors (RECIST 1.1), as assessed by blinded independent central review (BICR).
* Has received prior platinum-based chemotherapy and anti-programmed cell death 1 protein (PD-1)/anti- programmed cell death ligand 1 (PD-L1) therapy, either separately or in combination.

Exclusion Criteria:

* Has neuroendocrine tumors or endometrial sarcoma, including stromal sarcoma, leiomyosarcoma, adenosarcoma, or other types of pure sarcomas
* Has a history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has had a recurrence of endometrial carcinoma or carcinosarcoma more than >12 months after completing platinum-based therapy administered in the curative-intent setting without any additional platinum-based therapy received in the recurrent setting. Note: 1) If Immunotherapy-based treatment is administered in the recurrent setting, then platinum rechallenge is not required, regardless of the duration of the platinum-free interval from time of adjuvant therapy 2) For Stage IVb disease, treatment that includes gynecological surgery followed by a platinum-based regimen is NOT considered curative-intent per protocol and does not require platinum rechallenge in the recurrent setting, regardless of the duration of the platinum-free interval
* Has received more than 3 prior lines of therapy for endometrial carcinoma or carcinosarcoma
* Has history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has received prior treatment with single-agent nonplatinum based chemotherapy in the third-line setting
* Has received prior treatment with a trophoblast cell surface antigen 2 (TROP2)-targeted antibody drug conjugate (ADC) (eg, sacituzumab govitecan)
* Has received prior treatment with a topoisomerase I inhibitor-containing ADC (eg, sacituzumab govitecan or fam-trastuzumab deruxtecan-nxki)
* Has previously received both single-agent paclitaxel and single-agent doxorubicin in any setting for prior treatment of endometrial cancer
* Requires recurrent drainage of effusions (e.g., pleural, ascitic, etc.) within 6 weeks before randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2028-01-10 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 4 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 4 years
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 as Assessed by BICR | Up to approximately 4 years
  ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. based on BICR.
Duration of Response (DOR) per RECIST 1.1 as Assessed by BICR | Up to approximately 4 years
  For participants who demonstrate confirmed CR or PR per RECIST 1.1 as assessed by BICR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 4 years
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 4 years
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention whether or not considered related to the study intervention.
Change from Baseline in Global Health Status/Quality of Life Score (European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 [EORTC QLQ-C30]) | Baseline, up to approximately 4 years
  The EORTC QLQ-C30 is a questionnaire to assess the overall health status and quality of life of cancer patients. Participant responses to the questions, "How would you rate your overall health during the past week (Item 29)?" and "How would you rate your overall quality of life during the past week (Item 30)?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status and quality of life. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (241):
- United States (42):
  - USA Mitchell Cancer Institute ( Site 4142), Mobile, Alabama
  - Alaska Womens Cancer Care ( Site 4122), Anchorage, Alaska
  - HonorHealth (HH) ( Site 8000), Phoenix, Arizona
  - Arizona Oncology Associates - HOPE ( Site 8002), Tucson, Arizona
  - UCLA Hematology/Oncology - Westwood (Building 100)-Department of OBGYN, Division of Gynecologic Onc ( Site 4131), Los Angeles, California
  - California Pacific Medical Center - Van Ness Campus ( Site 4129), San Francisco, California
  - Yale-New Haven Hospital-Smilow Cancer Hospital at Yale-New Haven ( Site 4114), New Haven, Connecticut
  - MedStar Washington Hospital Center ( Site 4108), Washington D.C., District of Columbia
  - Mount Sinai Cancer Center ( Site 4117), Miami Beach, Florida
  - AdventHealth Orlando-AdventHealth Medical Group Gynecological Oncology ( Site 4113), Orlando, Florida
  - Florida Cancer Specialists - East ( Site 7000), West Palm Beach, Florida
  - Northside Hospital ( Site 4112), Atlanta, Georgia
  - Augusta University ( Site 4116), Augusta, Georgia
  - Centricity Research Columbus Cancer Center ( Site 4154), Columbus, Georgia
  - NorthShore University HealthSystem - Evanston Hospital ( Site 4110), Evanston, Illinois
  - Parkview Research Center at Parkview Regional Medical Center ( Site 4132), Fort Wayne, Indiana
  - Saint Elizabeth Medical Center Edgewood-Cancer Care Center ( Site 4150), Edgewood, Kentucky
  - University Medical Center New Orleans ( Site 4133), New Orleans, Louisiana
  - TRIALS 365 ( Site 4105), Shreveport, Louisiana
  - University of Massachusetts Memorial Medical Center ( Site 4103), Worcester, Massachusetts
  - Washington University School of Medicine-Obstetrics & Gynecology ( Site 4146), St Louis, Missouri
  - The Center of Hope ( Site 4109), Reno, Nevada
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 4118), Hackensack, New Jersey
  - Atlantic Health System Morristown Medical Center ( Site 4135), Morristown, New Jersey
  - Holy Name Medical Center ( Site 4115), Teaneck, New Jersey
  - New York - Presbyterian Brooklyn Methodist Hospital ( Site 4134), Brooklyn, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 4156), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center ( Site 4106), New York, New York
  - Icahn School of Medicine at Mount Sinai-Department of Obstetrics, Gynecology, and Reproductive Scie ( Site 4128), New York, New York
  - Good Samaritan Hospital Medical Center ( Site 4139), West Islip, New York
  - Duke Cancer Institute ( Site 4120), Durham, North Carolina
  - Sanford Health Roger Maris Cancer Center ( Site 4158), Fargo, North Dakota
  - University of Cincinnati Medical Center ( Site 4136), Cincinnati, Ohio
  - Sidney Kimmel Cancer Center - Jefferson Health ( Site 4157), Philadelphia, Pennsylvania
  - AHN West Penn Hospital-Gynecologic Oncology ( Site 4111), Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion ( Site 4107), Willow Grove, Pennsylvania
  - Women & Infants Hospital ( Site 4138), Providence, Rhode Island
  - Sanford Cancer Center-Gynecologic Oncology ( Site 4121), Sioux Falls, South Dakota
  - The West Clinic, PLLC dba West Cancer Center ( Site 4102), Germantown, Tennessee
  - Houston Methodist Hospital-Obstetrics and Gynecology ( Site 4130), Houston, Texas
  - Texas Oncology - San Antonio ( Site 8005), San Antonio, Texas
  - Texas Oncology - Gulf Coast ( Site 8006), The Woodlands, Texas
- Argentina (7):
  - Hospital Británico de Buenos Aires-Oncology ( Site 1002), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Argentino de Diagnóstico y Tratamiento (IADT) ( Site 1008), Buenos Aires, Buenos Aires F.D.
  - Instituto Alexander Fleming-Alexander Fleming ( Site 1007), Buenos Aires, Buenos Aires F.D.
  - Hospital Aleman-Oncology ( Site 1001), Buenos Aires
  - Instituto de Oncología Angel H. Roffo ( Site 1003), Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC) ( Site 1004), Buenos Aires
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 1006), La Rioja
- Australia (5):
  - GenesisCare North Shore ( Site 1103), St Leonards, New South Wales
  - Blacktown Hospital ( Site 1101), Sydney, New South Wales
  - Royal Brisbane and Women's Hospital ( Site 1102), Brisbane, Queensland
  - Epworth Freemasons ( Site 1104), East Melbourne, Victoria
  - Frankston Hospital ( Site 1105), Frankston, Victoria
- Austria (2):
  - Medizinische Universitaet Innsbruck-Univ.-Klinik f. Gynäkologie und Geburtshilfe ( Site 1201), Innsbruck, Tyrol
  - Medizinische Universität Wien ( Site 1202), Vienna
- Belgium (5):
  - AZ Maria Middelares-IKG ( Site 1305), Ghent, Oost-Vlaanderen
  - UZ Gent-Medical oncology ( Site 1303), Ghent, Oost-Vlaanderen
  - UZ Leuven-Gynecologic Oncology ( Site 1301), Leuven, Vlaams-Brabant
  - AZ Delta vzw-Oncology ( Site 1302), Roeselare, West-Vlaanderen
  - CHU UCL Namur/Site Sainte Elisabeth-Trial Office ( Site 1304), Namur
- Brazil (9):
  - Hospital São Domingos ( Site 1365), São Luís, Maranhão
  - Centro Oncologico do Triangulo ( Site 1360), Uberlândia, Minas Gerais
  - Hospital Moinhos de Vento ( Site 1359), Porto Alegre, Rio Grande do Sul
  - Instituto Joinvilense de Hematologia e Oncologia ( Site 1353), Joinville, Santa Catarina
  - Instituto de Ensino e Pesquisa ( Site 1355), Sorocaba, São Paulo
  - Instituto de Educação, Pesquisa e Gestão em Saúde ( Site 1352), Rio de Janeiro
  - Hospital Samaritano De Sao Paulo ( Site 1367), São Paulo
  - A. C. Camargo Cancer Center ( Site 1351), São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino ( Site 1366), São Paulo
- Canada (8):
  - Arthur J.E. Child Comprehensive Cancer Centre ( Site 1413), Calgary, Alberta
  - Cross Cancer Institute ( Site 1414), Edmonton, Alberta
  - BC Cancer Vancouver ( Site 1415), Vancouver, British Columbia
  - Trillium Health Partners - Credit Valley Hospital ( Site 1410), Mississauga, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean ( Site 1408), Chicoutimi, Quebec
  - CIUSSS de l'Est-de-l'Île-de-Montréal ( Site 1405), Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal ( Site 1403), Montreal, Quebec
  - McGill University Health Centre ( Site 1404), Montreal, Quebec
- Chile (4):
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 1505), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 1503), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 1501), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 1504), Temuco, Región de la Araucanía
- China (30):
  - Second Affiliated hospital of Anhui Medical University-Oncology ( Site 1635), Hefei, Anhui
  - Beijing Obstetric and Gynecology Hospital ( Site 1653), Beijing, Beijing Municipality
  - Fujian Cancer Hospital-Gynecological Oncology Surgery ( Site 1627), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University-Obstetrics and gynecology department ( Site 1613), Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University ( Site 1634), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center ( Site 1604), Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College ( Site 1642), Shantou, Guangdong
  - Affiliated Hospital of Guangdong Medical University ( Site 1614), Zhanjiang, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital-Gynecological oncology ( Site 1622), Nanning, Guangxi
  - Hainan General Hospital ( Site 1636), Haikou, Hainan
  - Harbin Medical University Cancer Hospital-Gynecological Radiotherapy Department ( Site 1652), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 1618), Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University ( Site 1640), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 1621), Wuhan, Hubei
  - Hubei Cancer Hospital-Hubei Cancer Hospital ( Site 1607), Wuhan, Hubei
  - Xiangya Hospital Central South University-Gynecology ( Site 1603), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 1623), Changsha, Hunan
  - Nanjing First Hospital ( Site 1649), Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital-Oncology Department ( Site 1625), Nanchang, Jiangxi
  - LinYi Cancer Hospital-Gastrology department ( Site 1630), Linyi, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University ( Site 1617), Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital-Gynecology department ( Site 1626), Shanghai, Shanghai Municipality
  - West China Second University Hospital, Sichuan University ( Site 1602), Chengdu, Sichuan
  - Sichuan Cancer hospital-Oncology ( Site 1650), Chengdu, Sichuan
  - Xinjiang Medical University Cancer Hospital - Urumqi ( Site 1648), Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital-Gynecology Department ( Site 1641), Kunming, Yunnan
  - The Affiliated Women's Hospital of Zhejiang University-Obstetrics and Gynecology ( Site 1609), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital-Oncology ( Site 1601), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 1633), Linhai, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 1615), Wenzhou, Zhejiang
- Czechia (7):
  - Fakultní Nemocnice Brno-Gynekologicko-porodnicka klinika ( Site 1704), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava-Gynekologicko-porodnicka klinika ( Site 1703), Ostrava, Moravskoslezský kraj
  - Nemocnice AGEL Novy Jicin a.s.-Oddeleni radioterapie a onkologie ( Site 1706), Nový Jiín, Novy Jicin
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 1702), Olomouc, Olomoucký kraj
  - Fakultni nemocnice Kralovske Vinohrady ( Site 1707), Prague, Praha 10
  - Vseobecna fakultni nemocnice v Praze-Gynekologicko-porodnicka klinika 1.LF a VFN ( Site 1705), Prague, Praha 2
  - Fakultni nemocnice Bulovka-Gynekologicko-porodnicka klinika ( Site 1701), Prague, Praha 8
- Denmark (3):
  - Herlev and Gentofte Hospital-Department of Oncology ( Site 1801), Copenhagen, Capital Region
  - Rigshospitalet-Dept. of Oncology ( Site 1803), Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby ( Site 1802), Aarhus, Central Jutland
- Finland (4):
  - Kuopion Yliopistollinen Sairaala ( Site 1904), Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala ( Site 1901), Tampere, Pirkanmaa
  - Turku University Hospital-Department of Obstetrics and Gynecology ( Site 1903), Turku, Southwest Finland
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 1902), Helsinki, Uusimaa
- France (10):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest ( Site 2002), Bordeaux, Aquitaine
  - CENTRE LEON BERARD ( Site 2004), Lyon Cedex08, Auvergne-Rhône-Alpes
  - ROC37 ( Site 2010), Chambray-lès-Tours, Centre-Val de Loire
  - Centre Armoricain de Radiotherapie Imagerie medicale et Oncologie ( Site 2001), Plérin, Cotes-d Armor
  - CHU Besançon ( Site 2009), Besançon, Doubs
  - Institut Claudius Regaud ( Site 2006), Toulouse, Haute-Garonne
  - Centre Oscar Lambret ( Site 2007), Lille, Hauts-de-France
  - Institut Regional du Cancer Montpellier ( Site 2008), Montpellier, Herault
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer ( Site 2003), Rennes, Ille-et-Vilaine
  - Groupe Hospitalier Diaconesses Croix Saint Simon ( Site 2005), Paris
- Germany (8):
  - SLK-Kliniken Heilbronn ( Site 2107), Heilbronn, Baden-Wurttemberg
  - Universitätsmedizin Mannheim-Department of Obstetrics and Gynecology ( Site 2101), Mannheim, Baden-Wurttemberg
  - MVZ für Hämatologie und Onkologie Ravensburg GmbH - Studienzentrum ( Site 2110), Ravensburg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen ( Site 2111), Tübingen, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern-Klinik und Poliklinik für Frauenheilkunde und Geburtshi ( Site 2109), Munich, Bavaria
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung ( Site 2104), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Frauenheilkunde und Gebur ( Site 2103), Dresden, Saxony
  - Charité Campus Virchow-Klinikum ( Site 2102), Berlin
- Greece (4):
  - Agios Andreas Hospital Patras ( Site 2201), Pátrai, Achaia
  - Aretaieio Hospital Oncology Unit ( Site 2206), Athens, Attica
  - Metropolitan Hospital-2nd Oncology Dept ( Site 2202), Athens, Attica
  - Hygeia Hospital ( Site 2204), Marousi, Attica
- Ireland (3):
  - Cork University Hospital ( Site 2402), Cork
  - Mater Misericordiae University Hospital ( Site 2403), Dublin
  - St. James's Hospital-Cancer clinical trials office ( Site 2401), Dublin
- Israel (6):
  - Rambam Health Care Campus-Gyneco-oncology unit ( Site 2502), Haifa
  - Edith Wolfson Medical Center ( Site 2501), Holon
  - Shaare Zedek Medical Center ( Site 2503), Jerusalem
  - Rabin Medical Center ( Site 2505), Petah Tikva
  - Sheba Medical Center ( Site 2504), Ramat Gan
  - Sourasky Medical Center ( Site 2506), Tel Aviv
- Italy (14):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlin-SSD Oncologia medica Addarii ( Site 2603), Bologna, Emilia-Romagna
  - CRO-IRCCS ( Site 2609), Aviano, Friuli Venezia Giulia
  - AOU Policlinico Umberto I ( Site 2606), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Chirurgia Ginecologica ( Site 2605), Milan, Lombardy
  - Istituto Europeo di Oncologia IRCCS ( Site 2607), Milan, Lombardy
  - Istituto Clinico Humanitas-U.O di Oncologia medica ed Ematologia ( Site 2610), Rozzano, Milano
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'O-Day Hospital Oncologico Multidisciplin ( Site 2613), Candiolo, Torino
  - Instituto Tumori Giovanni Paolo II-ONCOLOGIA MEDICA ( Site 2604), Bari
  - Azienda Ospedaliera Spedali Civili di Brescia-Obstetrics anf gynecology ( Site 2611), Brescia
  - Humanitas San Pio X Hospital ( Site 2614), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-S.C. Oncologia Sperimentale Uro-Genitale ( Site 2602), Napoli
  - Arcispedale Santa Maria Nuova ( Site 2612), Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Ginecologia Oncologica ( Site 2601), Roma
  - Ospedale Mauriziano-Ginecologia e Ostetricia ( Site 2608), Torino
- Japan (18):
  - Aichi Cancer Center ( Site 2714), Nagoya, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center ( Site 2705), Matsuyama, Ehime
  - Ehime University Hospital ( Site 2709), Tōon, Ehime
  - Kurume University Hospital ( Site 2703), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 2708), Otashi, Gunma
  - Hokkaido University Hospital ( Site 2707), Sapporo, Hokkaido
  - University of Tsukuba Hospital ( Site 2713), Tsukuba, Ibaraki
  - Iwate Medical University Hospital ( Site 2712), Shiwa-gun, Iwate
  - Niigata Cancer Center Hospital ( Site 2701), Niigata, Niigata
  - Saitama Medical University International Medical Center ( Site 2710), Hidaka, Saitama
  - Shizuoka Cancer Center ( Site 2716), Sunto-gun,, Shizuoka
  - National Cancer Center Hospital ( Site 2715), Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 2706), Koto, Tokyo
  - Showa Medical University Hospital ( Site 2719), Shinagawa, Tokyo
  - Keio University Hospital ( Site 2702), Shinjuku, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 2711), Fukuoka
  - Kagoshima City Hospital ( Site 2717), Kagoshima
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 2718), Osaka
- Malaysia (2):
  - Pantai Hospital Kuala Lumpur-Cancer Centre ( Site 2803), Kuala Lumpur
  - University Malaya Medical Centre ( Site 2801), Kuala Lumpur
- Mexico (5):
  - COI Centro Oncologico Internacional S.A.P.I. de C.V. ( Site 2902), Coyoacán, Mexico City
  - Higiea Oncologia ( Site 2905), Mexico City, Mexico City
  - Oncare - Unidad Valle ( Site 2906), San Pedro Garza García, Nuevo León
  - CENTRO MEDICO ZAMBRANO HELLION-Centro de Cáncer de Mama ( Site 2901), San Pedro Garza García, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 2907), Oaxaca City, Oaxaca
- Netherlands (3):
  - Radboudumc-Medical Oncology ( Site 3003), Nijmegen, Gelderland
  - Amsterdam UMC - locatie VUmc ( Site 3004), Amsterdam, North Holland
  - Leids Universitair Medisch Centrum-Medical Oncology ( Site 3002), Leiden, South Holland
- Norway (4):
  - Stavanger Universitetssykehus ( Site 3103), Stavanger, Rogaland
  - Universitetssykehuset Nord-Norge HF ( Site 3101), Tromsø, Troms
  - Sorlandet Sykehus Kristiansand ( Site 3104), Kristiansand, Vest-Agder
  - Oslo universitetssykehus, Radiumhospitalet ( Site 3102), Oslo
- Poland (4):
  - Wielkopolskie Centrum Onkologii im. Marii Skłodowskiej-Curie-Oddział Radioterapii i Onkologii Ginek ( Site 3202), Poznan, Greater Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 3201), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Ginekologii Onkologicznej ( Site 3203), Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii-Oddzial Onkologii Ginekologicznej ( Site 3204), Bialystok, Podlaskie Voivodeship
- Puerto Rico (3):
  - Ad-Vance Medical Research-Research ( Site 3302), Ponce
  - Pan American Center for Oncology Trials - Ciudadela ( Site 3301), San Juan
  - UPR Comprehensive Cancer Center-Comprehensive Cancer Center Hospital ( Site 3304), San Juan
- National Cancer Centre Singapore-Medical Oncology ( Site 3401), Singapore, Central Singapore, Singapore
- South Korea (5):
  - Seoul National University Bundang Hospital-Obstetrics and Gynecology ( Site 3505), Seongnam, Kyonggi-do
  - Seoul National University Hospital ( Site 3502), Seoul
  - Severance Hospital, Yonsei University Health System-Gynecologic cancer center ( Site 3503), Seoul
  - Asan Medical Center-Division of Gynecologic Oncology, Dept. of Obstetrics & Gynecology ( Site 3501), Seoul
  - Samsung Medical Center ( Site 3504), Seoul
- Spain (9):
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 3608), L'Hospitalet de Llobregat, Barcelona
  - Institut Català d'Oncologia (ICO) - Girona-Oncología Médica ( Site 3606), Girona, Gerona
  - Clinica Universidad de Navarra ( Site 3603), Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre-Medical Oncology ( Site 3607), Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz-Oncología Médica ( Site 3604), Madrid, Madrid, Comunidad de
  - Fundación Instituto Valenciano de Oncología-Oncologico ( Site 3605), Valencia, Valenciana, Comunitat
  - HOSPITAL CLINICO DE VALENCIA ( Site 3609), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 3602), Barcelona
  - Hospital Universitario Reina Sofia-Oncologia Medica ( Site 3601), Córdoba
- Sweden (2):
  - Skånes Universitetssjukhus Lund ( Site 3702), Lund, Skåne County
  - Karolinska Universitetssjukhuset Solna ( Site 3701), Stockholm, Stockholm County
- Switzerland (4):
  - University Hospital Basel-Gynecology & Gynecologic Oncology ( Site 3808), Basel, Canton of Basel-City
  - Ospedale Regionale Bellinzona e Valli ( Site 3802), Bellinzona, Canton Ticino
  - Kantonsspital Graubünden-Medizin ( Site 3803), Chur, Kanton Graubünden
  - Inselspital Bern-Oncology ( Site 3801), Bern
- United Kingdom (10):
  - University Hospitals Sussex NHS Foundation Trust ( Site 4006), East Sussex, Brighton And Hove
  - Royal Derby Hospital ( Site 4007), Derby, Derbyshire
  - ROYAL MARSDEN HOSPITAL (CHELSEA)-Gynaecology Research Centre ( Site 4002), London, England
  - The Royal Cornwall Hospital ( Site 4009), Truro, England
  - University College London Hospital-Cancer Clinical Trials Unit ( Site 4004), London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust-Oncology & Haematology Clinical Trials ( Site 4008), London, London, City of
  - Hammersmith Hospital ( Site 4001), London, London, City of
  - The Beatson West of Scotland Cancer Centre ( Site 4005), Glasgow, Scotland
  - Royal Marsden Hospital (Sutton)-Gynaecology Unit ( Site 4010), London, Sutton
  - The Christie NHS Foundation Trust-Medical Oncology ( Site 4003), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26130&tenant=MT_MSD_9011